CLINICAL TRIAL: NCT01045681
Title: A Phase II Study of Bendamustine, Velcade and Dexamethasone (BVD) in the Treatment of Elderly Patients (>= 65 Years) With Multiple Myeloma in 1st Relapse or Refractory to 1st Line Therapy
Brief Title: Study of Bendamustine, Velcade and Dexamethasone in the Treatment of Elderly Patients With Multiple Myeloma
Acronym: BVD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFM2009-01; Eudract 2009-012359-91 (Registry Identifier: AFSSAPS)
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2012-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Elderly patients; first relapse; refractory to first line therapy; Bendamustine Velcade Dexamethasone Association
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BVD (Experimental): Bendamustine, Velcade and Dexamethasone
  Interventions: Drug: Bendamustine, Velcade and Dexamethasone

INTERVENTIONS:
Drug: Bendamustine, Velcade and Dexamethasone — Bendamustine : 70 mg/m2 iv on D1 and 8, for each cycle Velcade : 1.3 mg/m2 iv on D1, 8, 15 and 22, for each cycle Dexamethasone : 20 mg/day po on D1, 8, 15 and 22, given prior to Bendamustine and Velcade
  Other Names: Robimustin : Bendamustine; Velcade : Bortezomib; Dexamethasone

SUMMARY:
The present trial is designed as a phase II study that aims at estimating the efficacy of the combination of bendamustine, bortezomib and dexamethasone in relapsed/refractory multiple myeloma (MM). The response rate, i.e. the rate of the patients achieving a Complete Response or Partial Response at cycle 4, divided by the total intent to treat patient number is chosen as primary efficacy endpoint.

The estimation of the efficacy rate is to be based on an explorative pilot study, since immediate embarking on a large-scale comparative efficacy trial would not be acceptable from the point of view of resources. Moreover, this would induce ethical objections, as it does not seem to be justifiable to expose a large number of patients to an experimental approach without sufficient exploratory indications of an improved risk-benefit ratio.

DETAILED DESCRIPTION:
After relapse or after early progression on first-line treatment, the prognosis of multiple myeloma (MM) patients is unfavourable, and the search for new treatment regimens, including drugs with novel mechanisms of action is essential.

Bendamustine and bortezomib have shown high activity boch in first-line regimens and pre-treated patients. The novel mechanism of action of the proteasome inhibitor and the non-cross resistance of bendamustine to other alkylating agents established in the first-line treatment of multiple myeloma seem to recommend a combination of the two drugs for salvage therapy (second-line regimen). Finally, the promising response data in a series of relapsing MM patients treated with bendamustine, bortezomib and prednisone support this assumption, as well as the feasibility and tolerability of the combination.

In summary, there is some evidence for a favorable risk/benefit ratio for the combination of bendamustine, bortezomib and a corticoid drug, warranting the exploration in a larger, prospectively designed multicenter phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma (MM) patient at the time of diagnosis (but not necessarily at the time of relapse), according to International Myeloma Working Group criteria.
* Patient having received conventional chemotherapy in 1st line treatment because of age 65 years or over, or younger than 65 years and ineligible to high-dose therapy plus stem cell transplantation.
* Measurable disease (≥10g/L monoclonal gammapathy and/or ≥ 200 mg/24h proteinuria or involved serum free light chain ≥ 100mg/L with abnormal FLC ratio < 0.26 or > 1.65)
* Patient in 1st relapse or refractory to 1st line therapy. Relapse is defined by M-component increase of ≥25% from baseline, in serum and/or urine (the absolute increase in serum must be ≥ 5 g/l - the absolute increase of BJ proteins in urine must be ≥200 mg/24 h). (It is recommended to treat only symptomatic or rapidly evolutive relapses)
* Life expectancy of at least 3 months
* ECOG performance status <= 2 at study entry
* Laboratory test results within these ranges:
* Absolute neutrophil count >= 1.5 x 109/L
* Platelet count >= 100 x 109/L
* Serum creatinine <= 250 umol/l
* AST (SGOT) and ALT (SGPT) <= 3 x ULN
* Disease free of prior malignancies for >= 5 years, with exception of curatively treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* Able to adhere to the study visit schedule and other protocol requirements
* Using effective contraceptive methods during and for 6 months after study treatment (for fertile men, women of childbearing potential).
* Provision of informed consent.
* A period of at least 15 days must be respected between the last treatment of myeloma and the beginning of the study.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Any comorbidity which places the subject at unacceptable risk if he/she were to participate in the study.
* Patients treated with high-dose therapy plus stem cell transplantation in 1st line therapy
* Any prior use of bortezomib (Velcade) or bendamustine (Ribomustin)
* Concurrent use of other anti-cancer agents or treatments other than those stated in this treatment plan
* Use of any other experimental drug or therapy within 28 days prior to the start of study treatment.
* Known hypersensitivity to the study drugs
* Positive HIV serology, positive hepatitis C serology, active infection hepatitis A, active infection hepatitis B.
* Severe cardiovascular disorders within 12 months prior to the start of study treatment (e.g. myocardial infarct, ischemic episodes, arrhythmias)
* Previous major surgery less than 30 days before start of treatment
* Active infection,
* Pregnant or lactating women.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-03-03 (Actual); Primary Completion 2013-03-28 (Actual); Study Completion 2013-03-28 (Actual)

PRIMARY OUTCOMES:
To assess of the overall response rate (complete response (CR) + partial response (PR)) | After four 28-day consecutives cycles

SECONDARY OUTCOMES:
Time to best response | the time from treatment start to the first detection of the best response category, calculated for all patients, which are not primarily refractory
Progression-free survival | The time form the initial dose of chemotherapy to the time of disease progression or death, or to the date of last assessment without any such event (censored observation)
Time to progression | The time from baseline to the development of progressive disease
Overall survival | The time interval from initial dose to the date of death or last observation (censored)
Rate of additional response | Following 2 consolidation cycles and following 6 maintenance cycles
Toxicity/Adverse events | From the time a signed and dated informed consent form is obtained until 60 days following the lase dose of study medication or until the start of a new subsequent antimyeloma therapy

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RODON, Doctor, Principal Investigator — Unité Hématologie Biologique Institut Curie PARIS; Cyrille HULIN, Doctor, Principal Investigator — Service Hématologie Hôpitaux de Brabois VANDOEUVRE LES NANCY; Jean-Luc HAROUSSEAU, Professor, Study Director — Service Hématologie CHU Nantes; Claire MATHIOT, Doctor, Study Chair — IFM Hématologie Biologique Institut Curie PARIS; Marie-Odile PETILLON, Doctor, Study Chair — IFM Hôpital Claude Huriez Lille
Locations (37):
- France (37):
  - CHRU Hôpital Sud, Amiens
  - CHRU, Hôpital du Bocage, Angers
  - Centre Hospitalier H.Duffaut, Avignon
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Hôpital Jean Minjoz / CHU BESANCON, Besançon
  - Centre Hospitalier, Blois
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital A.Morvan, Brest
  - Centre F.Baclesse, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU DIJON, Hôpital Le Bocage, Dijon
  - Centre Hospitalier Général, Dunkirk
  - Hôpital A.Michallon, Grenoble
  - CH Départemental, La Roche-sur-Yon
  - Centre Hospitalier de Chartres, Le Coudray
  - Centre Jean Bernard, Le Mans
  - CHRU Hôpital Claude Huriez, Lille
  - Institut Paoli Calmette, Marseille
  - CH MEAUX, Meaux
  - CHRU Hôtel Dieu, Nantes
  - Hôpital de l'Archet 1, Nice
  - Intitut Curie, Paris
  - CHU Hôpital St-Antoine, Paris
  - Centre Hopsitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier René Dubos, Pontoise
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - CHU Reims Hôpital R.Debré, Reims
  - CHRU - Hôpital sud, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - CHRU Hopital Purpan, Toulouse
  - CHRU Hopital Bretonneau, Tours
  - Centre Hospitalier, Valence
  - CHRU - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - CH P.Chubert, Vannes

REFERENCES:
- [Derived] Rodon P, Hulin C, Pegourie B, Tiab M, Anglaret B, Benboubker L, Jardel H, Decaux O, Kolb B, Roussel M, Garderet L, Leleu X, Fitoussi O, Chaleteix C, Casassus P, Lenain P, Royer B, Banos A, Benramdane R, Cony-Makhoul P, Dib M, Fontan J, Stoppa AM, Traulle C, Vilque JP, Petillon MO, Mathiot C, Dejoie T, Avet-Loiseau H, Moreau P. Phase II study of bendamustine, bortezomib and dexamethasone as second-line treatment for elderly patients with multiple myeloma: the Intergroupe Francophone du Myelome 2009-01 trial. Haematologica. 2015 Feb;100(2):e56-9. doi: 10.3324/haematol.2014.110890. Epub 2014 Nov 14. No abstract available. PMID 25398832